CLINICAL TRIAL: NCT06021431
Title: Digital Therapeutic Development of Virtual Cognitive-Affective Training for Opioid Use Disorder: A Phase 2 Randomized Controlled Trial
Brief Title: Virtual Reality Cognitive-Affective Training for Opioid Use Disorder- A Phase 2 RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BehaVR LLC (Industry)
Collaborators: University of Utah (Other); National Institute on Drug Abuse (NIDA) (NIH); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00157860; 5R44DA053848 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder
Keywords: Mindfulness; Virtual Reality; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MORE-VR (Experimental): An 8-session version of Mindfulness-Oriented Recovery Enhancement (MORE) delivered by virtual reality. The treatment involves training in mindfulness, reappraisal, and savoring techniques to address OUD.
  Participants in this arm will also receive Treatment as usual (TAU) with medications for opioid use disorder (MOUD) such as buprenorphine, methadone, or naltrexone plus any psychological counseling they are already receiving in their standard care.
  Interventions: Device: MORE-VR; Other: Treatment as Usual
- Treatment as Usual (TAU) (Active Comparator): Treatment as usual (TAU) with medications for opioid use disorder (MOUD) such as buprenorphine, methadone, or naltrexone plus any psychological counseling they are already receiving in their standard care.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: MORE-VR — An 8-session version of Mindfulness-Oriented Recovery Enhancement (MORE) delivered by virtual reality. The treatment involves training in mindfulness,reappraisal, and savoring techniques to address OUD.
  Combination Product: Participants in this arm will also receive Treatment as usual (TAU) with medications for opioid use disorder (MOUD). Usual addictions treatment with medications such as buprenorphine or methadone plus psychological counseling.
  Other Names: Mindfulness-Oriented Recovery Enhancement in Virtual Reality
  Arms: MORE-VR
Other: Treatment as Usual — Participants will receive their usual treatment for OUD, including medications such as buprenorphine or methadone and any counseling they might already be receiving

SUMMARY:
The goal of this clinical trial is to examine the usefulness of a virtual reality-delivered intervention for individuals with opioid use disorder who are taking medication. The main question it aims to answer is will people with opioid use disorder who receive the study intervention, Mindfulness-Oriented Recovery Enhancement in Virtual Reality (MORE-VR), have fewer days in which they use opioids than will people who just receive their usual treatment. Participants will be randomly assigned to either receive 8 weekly sessions of MORE-VR in addition to their usual treatment, or treatment as usual only. Researchers will compare these groups at the end of treatment and three months after treatment is over on number of days of opioid use and time until first opioid use lapse, as well as drug craving and mood.

DETAILED DESCRIPTION:
This project is a Phase II, two-arm, parallel randomized controlled trial (RCT) of a virtual reality form of Mindfulness-Oriented Recovery Enhancement (MORE-VR) versus treatment as usual (TAU) for patients receiving medications for opioid use disorder (MOUD) to assess the efficacy of the MORE-VR system. Participants will be randomized (1:1) to either 8 weekly sessions of MORE-VR or TAU. Participants will be assessed at intake, post-treatment, and a 3 month post-treatment follow-up. The primary outcome assessed will be days of opioid use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* current DSM-5 OUD diagnosis
* prescribed medications for opioid use disorder (e.g., buprenorphine, methadone)

Exclusion Criteria:

* completion of a standardized mindfulness intervention (e.g., MORE, MBRP, MBSR)
* active psychosis or suicidality
* reports, or is noted by clinical or study staff as showing cognitive impairment
* condition which might be contraindicated for VR use including seizure disorder, vertigo, severe motion sickness, recent concussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Days of opioid use | Baseline to post-treatment assessment (8 weeks)
  Days of opioid use assessed with the Timeline Followback method, ecological momentary assessments, and/or drug toxicology screen

SECONDARY OUTCOMES:
Days of opioid use at follow-up | Baseline to 3 months post treatment (20 weeks from baseline)
  Days of opioid use assessed with the Timeline Followback method, ecological momentary assessments, and/or drug toxicology screen
Time until opioid lapse | Baseline through 3 month post-treatment follow-up
  Number of days until opioid lapse assessed with the Timeline Followback method, ecological momentary assessments, and/or drug toxicology screen
Time until dropout from opioid use disorder treatment | Baseline through 3 month post-treatment follow-up
  Number of days unti dropout from treatment, assessed by Timeline Followback and chart review
Desire for drugs | Baseline, post-treatment, 3 month post-treatment follow-up, and weekly during intervention period
  Desires for Drug Questionnaire, range from 14 to 98, higher scores indicating more intense desires for drugs
Opioid craving | Baseline, post-treatment, 3 month post-treatment follow-up, and weekly during intervention period
  0-10 numeric rating scale via ecological momentary assessment (0=no craving, 10=extreme craving).
Positive Affect | Baseline, post-treatment, 3 month post-treatment follow-up, and weekly during intervention period
  0-10 numeric rating scale via ecological momentary assessment (0=no positive affect, 10=extremely strong positive affect).
Negative Affect | Baseline, post-treatment, 3 month post-treatment follow-up, and weekly during intervention period
  0-10 numeric rating scale via ecological momentary assessment (0=no negative affect, 10=extremely strong negative affect).
Positive and Negative Affect Schedule | Baseline, post-treatment, 3 month post-treatment follow-up, and weekly during intervention period
  A 20-item scale measuring both positive and negative affect, where each affective term is rated on a scale of 1 (not at all) to 5 (very much)
Distress | Baseline through 3 month post-treatment follow-up
  Emotional distress measured by the Depression Anxiety Stress Scale, range from 0 to 63, higher scores indicating worse distress.
Health-related Quality of Life | Baseline through 3 month post-treatment follow-up
  World Health Organization Quality of Life Scale Quality of life measured by the World Health Organization Quality of Life Scale (WHO-5), scores ranging from 0 to 25, with higher scores indicating better quality of life.

OTHER OUTCOMES:
Drug cue reactivity | Baseline to immediately after the intervention
  For a subset of participants, we will asses change from baseline in neurophysiological response during lab-based task involving presentation of drug cues designed to measure cue-reactivity.
Emotion regulation | Baseline to immediately after the intervention
  For a subset of participants, we will assess change from baseline in neurophysiological response during lab-based task involving presentation of emotional stimuli.
Theta oscillations | Baseline to immediately after the intervention
  For a subset of participants, we will assess theta oscillations as measured by EEG during meditation

CONTACTS AND LOCATIONS:
Overall Officials: Risa Weisberg, PhD, Principal Investigator — BehaVR LLC
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication of the primary, secondary, and mechanistic outcomes of the trial.
Access Criteria: Data will be available with a signed data access agreement